CLINICAL TRIAL: NCT04084314
Title: Assessment of Prolonged Safety and tOLerability of in Migraine Patients in a Long-term OpeN-label Study
Acronym: APOLLON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CAMG334ADE03; 2019-002201-22 (EudraCT Number)
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Migraine; Migraine Disorders; Migraine Headache
Keywords: migraine; episodic migraine; chronic migraine; headache; erenumab; AMG334; aimovig; monoclonal antibody; CGRP-receptor antibody
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Erenumab (Experimental): Erenumab dose could be adjusted from 70 mg to 140 mg or vice versa at the discretion of the physician at any scheduled study visit.
  Interventions: Biological: Erenumab

INTERVENTIONS:
Biological: Erenumab — Erenumab was supplied as a pre-filled pen (auto-injector) for subcutaneous injection.
  Other Names: AMG334; Aimovig

SUMMARY:
This is a 128-week open-label study to assess the long-term safety and tolerabilty of the monoclonal antibody erenumab in migraine patients.

DETAILED DESCRIPTION:
This was an open-label, multi-center, single arm study with flexible dosing allowing both dose adjustment and one drug holiday per patient.

The study design consisted of 3 parts:

* Screening Epoch (0 - 2 weeks): required for all patients to assess initial eligibility. Eligible patients came from study CAMG334ADE01 (NCT03828539).
* Open-label Treatment Epoch (128 weeks): Individual patients were treated for 128 weeks. In this open-label treatment phase, the erenumab dose could be adjusted from 70 mg to 140 mg or vice versa at the discretion of the physician at any scheduled study visit. Additionally, a voluntary single treatment interruption ('drug holiday') of up to 24 weeks (approximately six months) could be introduced after at least 12 weeks of treatment in the open-label Treatment Epoch.
* Follow-up Epoch (4 weeks): A Follow-Up Visit 4 weeks after the last regular study visit (8 weeks after last investigational medicinal product [IMP] application) was required as part of routine safety monitoring.

ELIGIBILITY:
The study population consisted of patients with a documented history of episodic (4 - 14 baseline migraine days) or chronic migraine (≥15 baseline headache days), who had been successfully randomized to clinical trial CAMG334ADE01.

Key inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study
* Patient is capable of understanding the nature, significance and implications of the clinical trial.
* Adults ≥18 years of age upon entry into screening

Key exclusion Criteria:

* Use of a prophylactic migraine medication within five plasma clearance half-lives, or a device or procedure within one month prior to the start of the Open-label Treatment Epoch. This exclusion criteria does not apply to erenumab or topiramate administered within clinical trial CAMG334ADE01
* Any prior exposure to (investigational) prophylactic migraine products targeting the CGRP pathway, other than erenumab.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-03-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (61):
- Germany (61):
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Marburg Wehrda, Germany
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Aachen, North Rhine-Westphalia
  - Novartis Investigative Site, Alzenau in Unterfranken
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Bad Honnef
  - Novartis Investigative Site, Bad Saarow
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dillingen
  - Novartis Investigative Site, Erbach im Odenwald
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Gelsenkirchen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Haar
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Hoppegarten
  - Novartis Investigative Site, Ibbenbueren
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Jülich
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Königstein im Taunus
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lünen
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Mittweida
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neu-Ulm
  - Novartis Investigative Site, Neuburg an der Donau
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Pforzheim
  - Novartis Investigative Site, Quakenbrück
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rülzheim
  - Novartis Investigative Site, Schwerin
  - Novartis Investigative Site, Seesen
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Sindelfingen
  - Novartis Investigative Site, Stadtroda
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Unterhaching
  - Novartis Investigative Site, Westerstede Oldenburg
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Gobel H, Schlegel E, Jaeger K, Ortler S, Leist L. Assessment of prolonged safety and tolerability of erenumab in migraine patients in a long-term open-label study (APOLLON). J Headache Pain. 2024 Sep 25;25(1):157. doi: 10.1186/s10194-024-01860-w. PMID 39322961
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1901

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 79 investigative sites in Germany.
Pre-assignment Details: The screening period began once patients had signed the study informed consent. The Screening Epoch had a duration of 2 weeks. Eligible patients came from study CAMG334ADE01 (NCT03828539).
Period: Overall Study
Arm/Group | Erenumab
Started | 701
Completed (Study Completed) | 534
Not Completed | 167
Not completed — Subject/guardian decision | 91
Not completed — Adverse Event | 24
Not completed — Lost to Follow-up | 19
Not completed — New therapy for study indication | 9
Not completed — Pregnancy | 9
Not completed — Withdrawal of informed consent | 8
Not completed — Physician Decision | 4
Not completed — Protocol Deviation | 3

BASELINE CHARACTERISTICS:
Arm/Group | Erenumab
Number analyzed (Participants) | 701
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 608
  Male | 93
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 695
  Asian | 1
  Unknown | 1
  Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Exposure Adjusted Incidence Rate of AE During Open-label Treatment Epoch Per 100 Subject Years
Description: This outcome measure was calculated dividing the number of adverse events (AEs) by the total patient exposure time and standardizing it per 100 patient-years. Exact Pearson-Clopper confidence intervals for single proportions were calculated to evaluate the precision of the estimated parameter.
Time Frame: Up to 128 weeks
Population: Safety set (SAF) defined as all patients who received at least one dose of study treatment in the Open-label Treatment Epoch of this study.
Measure: Number (95% Confidence Interval); unit: number of AEs per 100 patient-years
Arm/Group | Erenumab
Number analyzed (Participants) | 701
number of AEs per 100 patient-years | 101.71 [92.28 to 111.14]

2. Secondary Outcome: Proportion of Patients Discontinuing Open-label Treatment Epoch Due to AE
Description: Participants discontinuing the Open-label Treatment Epoch due to adverse events (AEs) to evaluate the long-term tolerability of erenumab in patients with episodic migraine or chronic migraine.
Time Frame: Up to 128 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab
Number analyzed (Participants) | 701
Participants | 29

3. Secondary Outcome: Proportion of Patients Discontinuing Open-label Treatment Epoch Due to Non-AE Reasons
Description: Participants discontinuing the Open-label Treatment Epoch due to non-AE reasons to evaluate the long-term tolerability of erenumab in patients with episodic migraine or chronic migraine.
Time Frame: Up to 128 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab
Number analyzed (Participants) | 701
Participants | 126

ADVERSE EVENTS:
Time Frame: From first dose of study treatment in the Open-label Treatment Epoch of this study to 8 weeks after last dose (up to 132 weeks).
Arm/Group | Erenumab
All-Cause Mortality (participants affected / at risk) | 0/701
Serious Adverse Events (participants affected / at risk) | 86/701
Other Adverse Events (participants affected / at risk) | 514/701
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab (N=701)
Atrial fibrillation (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Macrocornea (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Vestibular paroxysmia (Ear and labyrinth disorders) | 1
Goitre (Endocrine disorders) | 1
Cataract (Eye disorders) | 1
Lens dislocation (Eye disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Internal hernia (Gastrointestinal disorders) | 1
Intestinal stenosis (Gastrointestinal disorders) | 1
Large intestinal stenosis (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Volvulus (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Capsular contracture associated with breast implant (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Hypersensitivity (Immune system disorders) | 1
Appendicitis (Infections and infestations) | 4
Appendicitis perforated (Infections and infestations) | 1
Bartholinitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastrointestinal viral infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Nephritis bacterial (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Root canal infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vestibular neuronitis (Infections and infestations) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 2
Bursa injury (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Shoulder fracture (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 7
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Sacral pain (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebellar atrophy (Nervous system disorders) | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 2
Multiple sclerosis (Nervous system disorders) | 1
Nerve compression (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Retroplacental haematoma (Pregnancy, puerperium and perinatal conditions) | 1
Depression (Psychiatric disorders) | 5
Depression suicidal (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 2
Ureterolithiasis (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 2
Ovarian cyst (Reproductive system and breast disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Raynaud's phenomenon (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab (N=701)
Vertigo (Ear and labyrinth disorders) | 25
Abdominal pain upper (Gastrointestinal disorders) | 15
Constipation (Gastrointestinal disorders) | 103
Diarrhoea (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 34
Chills (General disorders) | 20
Fatigue (General disorders) | 61
Pyrexia (General disorders) | 20
COVID-19 (Infections and infestations) | 242
Cystitis (Infections and infestations) | 23
Nasopharyngitis (Infections and infestations) | 134
Tonsillitis (Infections and infestations) | 18
Urinary tract infection (Infections and infestations) | 18
Immunisation reaction (Injury, poisoning and procedural complications) | 43
Post vaccination fever (Injury, poisoning and procedural complications) | 15
Procedural pain (Injury, poisoning and procedural complications) | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 33
Back pain (Musculoskeletal and connective tissue disorders) | 42
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29
Dizziness (Nervous system disorders) | 24
Headache (Nervous system disorders) | 42
Migraine (Nervous system disorders) | 43
Depression (Psychiatric disorders) | 39
Cough (Respiratory, thoracic and mediastinal disorders) | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20
Alopecia (Skin and subcutaneous tissue disorders) | 28
Pruritus (Skin and subcutaneous tissue disorders) | 18
Hypertension (Vascular disorders) | 46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT04084314/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT04084314/SAP_001.pdf